CLINICAL TRIAL: NCT06955364
Title: A New Measurement Tool for Investigation of Pain Monitoring and Post-Injury Effects in Athletes
Brief Title: Development Study of Pain Monitoring and Injury Impact Scale
Acronym: PAMIIS
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Şeyda ÖZAL, Principal Investigator (Master of Science degree Physiotherapist), Gazi University
Other Study IDs: GaziUnivrs
Record Dates: First submitted 2025-04-21; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Sports Injuries; Social Impact; Psychological Impact of Injury
Keywords: Pain monitoring; Scale development; Performance; Participation
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Pilot Study (pretest) Group: In the pilot study, the comprehensibility and feedback forms were administered to 30 athletes from various branches to assess the content and face validity of PAMIIS.
- Main Testing Group: The new version of PAMIIS was administered to 148 athletes for consistency and construct validity with Exploratory Factor Analysis (EFA). OSTRC-O and OSTRC-H questionnaires were also applied to investigate the concurrent validity of PAMIIS.
- Retest Group: The scale was reapplied to 55 athletes in the main test group one week later to check its reproducibility.
- Final Test Group: The remodeled PAMIIS was applied to the 90 athletes for Confirmatory Factor Analysis (CFA) of the PAMIIS to ensure its construct validity

SUMMARY:
This study introduced and validated the Pain Monitoring and Injury Impact Scale for Athletes (PAMIIS), developed to address the lack of a comprehensive tool in Turkish for assessing injury-related pain and its multidimensional impact on athletes.The development process involved expert consultations, literature review, and feedback from athletes, resulting in a 37-item pool that was refined through pilot testing. Psychometric analyses conducted with 148 athletes demonstrated strong internal consistency, high test-retest reliability, and substantial correlations with established tools such as the Visual Analog Scale, OSTRC-O, and OSTRC-H. The final scale structure, consisting of 32 items across four subscales, was confirmed through both exploratory and confirmatory factor analyses. PAMIIS is a psychometrically sound instrument for systematically monitoring athletes' health status and documenting the short- and long-term consequences of sports injuries.

DETAILED DESCRIPTION:
ABSTRACT Aims: In Turkish, there is no valid and reliable measurement tool for monitoring the health status of athletes and evaluating the effects of injuries on them from various dimensions. With this study, we aimed to develop a measurement tool to detect pain associated with sports injuries and to investigate the consequences of injury. We created a measurement tool called Pain Monitoring and Injury Impact Scale for Athletes-PAMIIS, which consists of a Pain Detection Diagram and an Injury Impact Scale.

Methods: PAMIIS was designed and improved upon expert, partner, and participant opinions and a literature review. Initially, a pool of 37 items was created. The content and scope of the tool were checked with a pilot test on 30 athletes. In the main test phase, 148 participants (200 sample) were tested for item consistency, and 55 athletes (70 sample) were retested for stability to determine reliability. For concurrent validity, PAMIIS sub-scores were compared with the Visual Analog Scale, the Oslo Sports Trauma Research Center Overuse Injury Questionnaire (OSTRC-O), and the Oslo Sports Trauma Research Center on Health Problems (OSTRC-H) scores. Scale structure revealed with Exploratory Factor Analysis (EFA) for the construct validity. In the final phase, 90 (122 sample) athletes were administered the restructured scale, and its construct was tested with Confirmatory Factor Analysis (CFA).

ELIGIBILITY:
Inclusion Criteria:

* Engaged in regular participation in any form of sporting activity for a minimum duration of six months
* Aged 13 years or older
* Had sufficient proficiency in the Turkish language to comprehend and respond to the study materials
* Voluntarily agreed to participate in the study, with informed consent obtained

Exclusion Criteria:

* Pregnancy or illiteracy

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All athletes who regularly participate in a sporting activity for more than six months, aged 13 or over, and Turkish-speaking.
Sampling Method: Probability Sample
Enrollment: 268 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Pain Monitoring and Injury Impact Scale (PAMIIS) | Baseline
  It is a two-tiered, self-reported scale designed to determine the health level of athletes through pain symptoms in all body parts and to investigate the physical, psychological, and social effects of injury on the athlete. The first tier of the scale includes a diagram that enables health monitoring and screening for athletes. This section involves querying the athlete about the presence of pain, if any, its localization, intensity, onset, progression, and its relationship with training. This section is designed to be repeated weekly in pain-free athletes to monitor changes in their condition. If the athlete is already injured or a painful condition is detected in the first tier, he is prompted to proceed to the second tier. Here, the Performance, Participation, Psychological, and Social impacts resulting from the injury are thoroughly investigated. An athlete gets a minimum of 0 and a maximum of 128 points on the injury impact scale. Higher points show worse health conditions.

SECONDARY OUTCOMES:
Oslo Sports Trauma Research Centre Questionnaires for Overuse Injury (OSTRC-O) | Baseline
  The "Oslo Sports Trauma Research Centre Questionnaires for Overuse Injury" is a self-reported outcome measure. It queries sports participation, training volume, sports performance, and pain for a selected body location-e.g. knee taking into account the last seven days. A severity score is between 0-100 points. Higher points show worse health conditions.
Oslo Sports Trauma Research Centre questionnaires on Health Problems (OSTRC-H) | Baseline
  "Oslo Sports Trauma Research Centre questionnaires on Health Problems" is a self-reported outcome measure. It is applied to determine the effects of general health problems on sports participation, training volume, sports performance, and pain for the last seven days. A severity score is between 0 and 100 points. Higher points show worse health conditions
Pain Monitoring and Injury Impact Scale (PAMIIS) | one week later
  It is a two-tiered, self-reported scale designed to determine the health level of athletes through pain symptoms in all body parts and to investigate the physical, psychological, and social effects of injury on the athlete. The first tier of the scale includes a diagram that enables health monitoring and screening for athletes. This section involves querying the athlete about the presence of pain, if any, its localization, intensity, onset, progression, and its relationship with training. This section is designed to be repeated weekly in pain-free athletes to monitor changes in their condition. If the athlete is already injured or a painful condition is detected in the first tier, he is prompted to proceed to the second tier. Here, the Performance, Participation, Psychological, and Social impacts resulting from the injury are thoroughly investigated. An athlete gets a minimum of 0 and a maximum of 128 points on the injury impact scale. Higher points show worse health conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Şeyda YILMAZ ÖZAL, Assistant Professor, Principal Investigator — Ankara Medipol University; Nihan KARATAŞ, Professor, Study Director — Gazi University; Nevin ATALAY GÜZEL, Professor, Study Chair — Gazi University; Melek Gülşah ŞAHİN, Professor, Study Chair — Gazi University
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara Medipol University, Ankara, Çankaya
  - Gazi University, Ankara, Çankaya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maffulli N, Longo UG, Gougoulias N, Caine D, Denaro V. Sport injuries: a review of outcomes. Br Med Bull. 2011;97:47-80. doi: 10.1093/bmb/ldq026. Epub 2010 Aug 14. PMID 20710023
- [Background] Meeuwisse WH. Assessing causation in sport injury: a multifactorial model. LWW; 1994. p. 166-170.
- [Background] Özal Ş, Kafa N, Güzel NA, Development of a measurement tool for investigation of pain monitoring and post-injury effects in athletes, Gazi University Institute of the Health Science PhD thesis 2023/4
- [Background] Yilmaz Ozal S, Kafa N, Yuksel F, Guzel N. Turkish translation and validation of the Oslo Sports Trauma Research Center (OSTRC) Questionnaires. Malawi Med J. 2025 Apr 2;37(1):44-50. doi: 10.4314/mmj.v37i1.7. eCollection 2025 Mar. PMID 41306359